CLINICAL TRIAL: NCT06943820
Title: A Phase Ib/II Study of Anti-PD-1/LAG-3 Bispecific Antibody AK129 Combinations in Advanced Solid Tumors
Brief Title: AK129 Combination Therapy for Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK129-201
Record Dates: First submitted 2025-04-06; First posted 2025-04-24 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Non-small Cell Lung Cancer Stage IIIB/IV; Head and Neck Squamous Cell Carcinoma (HNSCC); Colorectal Adenocarcinoma; Advanced Solid Tumors
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Pemetrexed; Paclitaxel; Carboplatin; Docetaxel; Cisplatin; Fluorouracil; Cetuximab; Drug Therapy; penpulimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- AK129(dose 1) + Chemotherapy(Phase Ib) (Experimental): Non-Squamous NSCLC:Subjects receive AK129 (dose 1) plus Pemetrexed and Carboplatin on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by AK129(dose 1) plus Pemetrexed until progression.
  Squamous NSCLC:Subjects receive AK129 (dose 1) plus Paclitaxel and Carboplatin on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by AK129(dose 1) until progression.
  Interventions: Drug: AK129(dose 1); Drug: Pemetrexed; Drug: Paclitaxel; Drug: Carboplatin
- AK129(dose 2) + Chemotherapy(Phase Ib) (Experimental): Non-Squamous NSCLC:Subjects receive AK129 (dose 2) plus Pemetrexed and Carboplatin on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by AK129(dose 2) plus Pemetrexed until progression.
  Squamous NSCLC:Subjects receive AK129(dose 2) plus Paclitaxel and Carboplatin on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by AK129(dose 2) until progression.
  Interventions: Drug: Pemetrexed; Drug: Paclitaxel; Drug: Carboplatin; Drug: AK129(dose 2)
- Cohort 1 PARTA Treatment Group 1(Phase II) (Experimental): Non-Squamous NSCLC:Subjects receive AK129 (RP2D) plus Pemetrexed and Carboplatin on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by AK129(RP2D) plus Pemetrexed until progression.
  Squamous NSCLC:Subjects receive AK129(RP2D) plus Paclitaxel and Carboplatin on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by AK129(RP2D) until progression.
  Interventions: Drug: Pemetrexed; Drug: Paclitaxel; Drug: Carboplatin; Drug: AK129(RP2D)
- Cohort 1 PARTA Treatment Group 2(Phase II) (Active Comparator): Non-Squamous NSCLC:Subjects receive Penpulimab plus Pemetrexed and Carboplatin on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by Penpulimab plus Pemetrexed until progression.
  Squamous NSCLC:Subjects receive Penpulimab plus Paclitaxel and Carboplatin on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by Penpulimab until progression.
  Interventions: Drug: Pemetrexed; Drug: Paclitaxel; Drug: Carboplatin; Drug: Penpulimab
- Cohort 1 PARTB(Phase II) (Experimental): NSCLC:Subjects receive AK129(RP2D) plus Docetaxel on Day 1 of every 3-week cycle (Q3W) until progression.
  Interventions: Drug: Docetaxel; Drug: AK129(RP2D)
- Cohort 2 PARTA(Phase II) (Experimental): HNSCC:Subjects receive AK129(RP2D,Day1) plus Carboplatin/Cis-platinum(Day1) and 5-FU(Day1-4) every 3-week cycle (Q3W) for 6 cycles followed by AK129(RP2D) until progression.
  Interventions: Drug: Carboplatin; Drug: Cis-platinum; Drug: 5-FU (5-fluorouracil); Drug: AK129(RP2D)
- Cohort 2 PARTB(Phase II) (Experimental): HNSCC:Subjects receive AK129(RP2D) plus 1 investigator-selected treatment protocol(Cetuximab/Paclitaxel/Docetaxel) on Day 1 of every 3-week cycle (Q3W) until progression, and are not allowed to choose a treatment they had already received.
  Interventions: Drug: Cetuximab; Drug: Paclitaxel; Drug: Docetaxel; Drug: AK129(RP2D)
- Cohort 3(Phase II) (Experimental): CRC:Subjects receive AK129(RP2D) until progression.
  Interventions: Drug: AK129(RP2D)
- Cohort 4(Phase II) (Experimental): Advanced solid tumors:Subjects receive AK129(RP2D)± chemotherapy until progression.
  Interventions: Drug: Chemotherapy; Drug: AK129(RP2D)

INTERVENTIONS:
Drug: AK129(dose 1) — IV infusion
  Arms: AK129(dose 1) + Chemotherapy(Phase Ib)
Drug: Pemetrexed — IV infusion;500mg/m2
  Arms: AK129(dose 1) + Chemotherapy(Phase Ib); AK129(dose 2) + Chemotherapy(Phase Ib); Cohort 1 PARTA Treatment Group 1(Phase II); Cohort 1 PARTA Treatment Group 2(Phase II)
Drug: Paclitaxel — IV infusion;175mg/m2
  Arms: AK129(dose 1) + Chemotherapy(Phase Ib); AK129(dose 2) + Chemotherapy(Phase Ib); Cohort 1 PARTA Treatment Group 1(Phase II); Cohort 1 PARTA Treatment Group 2(Phase II)
Drug: Carboplatin — IV infusion;AUC 5
  Arms: AK129(dose 1) + Chemotherapy(Phase Ib); AK129(dose 2) + Chemotherapy(Phase Ib); Cohort 1 PARTA Treatment Group 1(Phase II); Cohort 1 PARTA Treatment Group 2(Phase II); Cohort 2 PARTA(Phase II)
Drug: AK129(dose 2) — IV infusion
  Arms: AK129(dose 2) + Chemotherapy(Phase Ib)
Drug: Docetaxel — IV infusion;75mg/m2
  Arms: Cohort 1 PARTB(Phase II)
Drug: Cis-platinum — IV infusion;100 mg/m2
  Arms: Cohort 2 PARTA(Phase II)
Drug: 5-FU (5-fluorouracil) — IV infusion;1000 mg/m2
  Arms: Cohort 2 PARTA(Phase II)
Drug: Cetuximab — IV infusion;400mg/m2/ 250mg/m2
  Arms: Cohort 2 PARTB(Phase II)
Drug: Paclitaxel — IV infusion;80mg/m2
  Arms: Cohort 2 PARTB(Phase II)
Drug: Docetaxel — IV infusion;35mg/m2
  Arms: Cohort 2 PARTB(Phase II)
Drug: Chemotherapy — IV infusion
  Arms: Cohort 4(Phase II)
Drug: AK129(RP2D) — IV infusion
  Arms: Cohort 1 PARTA Treatment Group 1(Phase II); Cohort 1 PARTB(Phase II); Cohort 2 PARTA(Phase II); Cohort 2 PARTB(Phase II); Cohort 3(Phase II); Cohort 4(Phase II)
Drug: Penpulimab — IV infusion;200mg
  Arms: Cohort 1 PARTA Treatment Group 2(Phase II)

SUMMARY:
This is an open, multicenter phase Ib/II clinical study. The goal of this study is to confirm the Phase II recommended dose (RP2D) of AK129 combinations for advanced solid tumors and evaluate the safety and efficacy of AK129 combinations for non-small cell lung cancer (NSCLC), head and neck squamous cell carcinoma (HNSCC), colorectal adenocarcinoma (CRC), and other advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Be able and willing to provide written informed consent and to comply with all requirements of study participation (including all study procedures);
2. ≥18 years old and ≤ 75 years (regardless of sex);
3. ECOG performance status 0-1;
4. Life expectancy longer than 3 months;
5. 1)Histologically or cytologically confirmed diagnosis of Stage IIIB/C or IV NSCLC (American Joint Committee on Cancer [AJCC]); 2)No prior systemic anti-tumor therapy for locally advanced or metastatic NSCLC;must have received a platinum-based combination therapy and a PD-(L)1 monoclonal antibody for the treatment of locally advanced or metastatic disease and progressed during or after receiving prior therapy;
6. 1)Histologically or cytologically confirmed diagnosis of recurrent or metastatic HNSCC (American Joint Committee on Cancer [AJCC]); 2)No prior systemic anti-tumor therapy for recurrent or metastatic HNSCC ;must have received a platinum-based combination therapy and a PD-(L)1 monoclonal antibody for the treatment of recurrent or metastatic disease and progressed during or after receiving prior therapy;
7. Histologically or cytologically confirmed diagnosis of advanced colorectal adenocarcinoma with microsatellite stabilization;
8. Measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1;
9. Adequate organ function.

Exclusion Criteria:

1. Histologically or cytologically confirmed the presence of small cell carcinoma components/EGFR-sensitive mutations or ALK fusion positivite/known ROS1 rearrangement, MET exon 14 skipping mutation, EGFR exon 20 insertion mutation, BRAF V600E mutation, NTRK gene fusion positivite or RET gene fusion positivite;
2. Histologically or cytologically confirmed diagnosis of advanced colorectal adenocarcinoma with microsatellite highly unstable/mismatch repair gene expression defect (MSI-H/dMMR)or histopathological examination confirmed other pathological types;
3. Participating in another clinical research;
4. Has known active central nervous system (CNS) metastases, brain stem/meningeal metastasis, spinal cord metastasis or compression;
5. Has an active autoimmune disease that has required systemic treatment in the past 2 years;
6. Has known active tuberculosis (TB) and suspected active TB should be ruled out by clinical examination; known active syphilis infection; known active Hepatitis B or Hepatitis C;
7. Past or currently has non-infectious pneumonia/interstitial lung disease that requires systemic glucocorticoid therapy;
8. Has pleural effusion, pericardial effusion, or ascites that have clinical symptoms or require repeated drainage;
9. Had a history of myocarditis, cardiomyopathy, and malignant arrhythmia;
10. Has known allergy to any component of any investigational drug; a known history of severe hypersensitivity to other monoclonal antibodies;
11. Pregnant or lactating female.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events (AEs) ,Clinically significant abnormal laboratory results | Up to approximately 2 years
  Frequency and severity of AEs and clinically significant abnormal laboratory results for all arms in phase Ib/II.
Overall Response Rate (ORR) | Up to approximately 2 years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) for all arms in phase II , based on RECIST v1.1.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 2 years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) for all arms in phase Ib, based on RECIST v1.1.
Progression-Free Survival (PFS) | Up to approximately 2 years
  Evaluation of PFS based on RECIST v1.1.
Overall survival (OS) | Up to approximately 2 years
  Evaluation of OS based on RECIST v1.1.
Disease control rate (DCR) | Up to approximately 2 years
  Evaluation of DCR based on RECIST v1.1.
Duration of Response (DoR) | Up to approximately 2 years
  Evaluation of DoR based on RECIST v1.1.
Time to Response (TTR) | Up to approximately 2 years
  Evaluation of TTR based on RECIST v1.1.
Pharmacokinetics (PK) | Up to cycle 21(each cycle is 21 days)
  PK parameters: serum concentrations of AK129 at different point of time
Anti-Drug Antibodies(ADAs) | Up to approximately 2 years
  Number and percentage of patients with detectable anti-drug antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- Liaoning Cancer Hospital, Shenyang, Liaoning, China